CLINICAL TRIAL: NCT05407987
Title: Feasibility and Efficacy of Intravenous Ferric Derisomaltose to Correct Pre-operative Iron-deficiency Anemia in Patients Undergoing Gynecologic Oncology Surgery: a Pilot Randomized Double Blinded Parallel Group Placebo-controlled Study
Brief Title: Ferric Derisomaltose and Outcomes in the Recovery of Gynecologic Oncology: ERAS (Enhanced Recovery After Surgery)
Acronym: FORGE II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FORGE II
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Gynecologic Cancer; Anemia; Iron-deficiency
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency | interventions — ferric derisomaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Therapy Arm (Experimental): 500 or 1000mg of IV Ferric Derisomaltose in 100mL normal saline will be administered intravenously over 1 hour. Participants with bodyweight <50kg will receive 500mg, participants with bodyweight >50kg will receive 1000mg to ensure no patient exceeds the manufacturer's recommended dose of 20mg/kg bodyweight.
  Interventions: Drug: Ferric derisomaltose
- Placebo Arm (Placebo Comparator): 100mL of normal saline will be administered intravenously over 1 hour between 21 and 90 days preceding surgical intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric derisomaltose — Ferric Derisomaltose is a solution based iron supplement provided in 100 mg elemental iron/mL. Patients randomized to Iron Therapy Arm will with a bodyweight <50kg will receive 500mg of Ferric Derisomaltose, and patients with a bodyweight >50kg will receive 1000mg of Ferric Derisomaltose, to ensure no patient exceeds the manufacturer's recommended dose of 20mg/kg. Patients will receive a single infusion between 21 and 90 days preceding surgical intervention.
  Other Names: MONOFERRIC
  Arms: Iron Therapy Arm
Drug: Placebo — Patients randomized to the Placebo arm will receive 100mg of normal saline over 1 hour.
  Arms: Placebo Arm

SUMMARY:
Iron deficiency has been reported in approximately 35% of patients with a gynecologic malignancy. Blood transfusions are known to be immunosuppressive and carry immediate and long-term risks. Pre-operative blood transfusion in gynecologic oncology patients is associated with higher rates of surgical site infection, length of stay, composite morbidity, cancer recurrence, and mortality. Pre-operative intravenous iron formulations have been shown in benign gynecology and other surgical specialities to increase pre-operative hemoglobin and decrease post-operative transfusion rates.

This is a randomized double-blinded clinical trial evaluating the effects of treating patients undergoing gynecologic oncology surgery with intravenous ferric derisomaltose to correct pre-operative iron-deficiency anemia.

The study aims to assess the effectiveness of preoperative ferric derisomaltose/iron isomaltoside compared to placebo in correcting preoperative hemoglobin in patients undergoing surgery for gynecologic malignancy.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to initiation of any study specific activities/procedures.
2. Age ≥ 18 years old.
3. Patients undergoing elective major surgery on the gynecologic oncology service with the following criteria will be considered for inclusion:

   1. The indication for the operation may be for suspected or proven gynecologic malignancy.
   2. Major surgery is defined as an operation of a duration of 1 hour or greater, with an Aletti complexity score of at least 1.
   3. The expected time from recruitment to surgery is 28-90 days.
4. Screening haemoglobin less than 120 g/L and transferrin saturation (TSAT) <20%.
5. Randomization and administration of study infusion a minimum of 21 days and maximum 90 days before planned operation.
6. Negative pregnancy test for women of childbearing potential (WOCBP) (within 7 days prior to treatment).
7. WOCBP must adhere to the contraception requirement from screening throughout the study period until 6 weeks post treatment.
8. Laboratory data used for determination of eligibility (Hemoglobin and Transferrin saturation) at the baseline visit must not be older than 4 weeks.

Exclusion Criteria:

1. Known history of acquired iron overload, or family history of haemochromatosis or thalassemia, or TSAT >50%.
2. Known alternative cause for anemia (e.g., B12 or folate deficiency, or haemoglobinopathy).
3. Known hypersensitivity to Ferric derisomaltose/iron isomaltoside (Monoferric®) or its excipients.
4. Temperature >38C or patient on non-prophylactic antibiotics.
5. Known chronic liver disease or active hepatitis.
6. Received erythropoietin or IV iron therapy within previous 12 weeks prior to planned study drug treatment.
7. Alanine transaminase (ALT) or aspartate transaminase (AST) above three times the upper limit of normal (ULN) range.
8. Immunosuppressive therapy (for solid organ transplant), or renal dialysis (current, or planned within next 12 months following treatment with study drug or placebo).
9. Unfit for elective surgery.
10. Pregnancy or lactation.

1. Unable to fully comprehend and/or perform study procedures and patients with psychiatric illness/social situations/substance abuse that would limit compliance with study requirements.

11. Cervical cancer with a clinical stage of 2A or greater.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean preoperative haemoglobin concentration | Haemoglobin concentration will be measured at baseline and 3 days prior to surgery after treatment with Ferric Derisomaltose
  To determine the effect of IV iron supplementation provided at least 21 days prior to surgery for gynecologic malignancy on mean preoperative haemoglobin concentration (in g/L)in patients with iron deficiency anemia compared to those patients without preoperative IV iron supplementation.

SECONDARY OUTCOMES:
Mean haemoglobin concentration at the time of surgery | Haemoglobin concentration will be measured at baseline and at the time of surgery after treatment with Ferric Derisomaltose
  The effect of IV iron supplementation provided prior to surgery for gynecologic malignancy on mean haemoglobin concentration (in g/L) at the time of surgery.
Mean postoperative haemoglobin concentration | Haemoglobin concentration will be measured at 28 and 60 days after surgery
  The effect of IV iron supplementation provided prior to surgery for gynecologic malignancy on mean hemoglobin concentration after the completion of surgery which will be assessed by measuring blood hemoglobin levels
Assessment of the requirement of postoperative blood transfusion | Day 0 to 28 days following surgery
  The number of participants requiring blood transfusion after completion of gynecologic surgery. A blood transfusion event is defined as receiving any volume of one unit or more than one unit of packed red cells or whole blood.
Mean number of blood transfusions | Day 0 to 28 days following surgery
  The mean number of blood transfusion (total number of units of packed red blood cells transfused ) after completion of gynecologic surgery
Postoperative Quality of Recovery(QoR)-15 questionnaire score | Post-operation day 1 (24 hours ± 12 hours following surgery)
  Quality of life will be evaluated using Quality of Recovery(QoR)-15 questionnaire score at postoperative day 1 compared to baseline (minimum value : 0, maximum value : 150, the higher the score, the better the result)
Mean Change in the Functional Assessment of Cancer Therapy-Anemia (FACT-An) Scores | Baseline to 0-3 days prior to surgery and at 23-33 days postoperative
  The FACT-An questionnaire is a 47-item, cancer specific questionnaire consisting of a core 27 items measuring 4 general domains physical well being (PWG), social/family (SWB), emotional well being (EWB) and Functional Well-Being (FWB) and an additional 20-item anemia questionnaire that measures fatigue associated items and 7 non-fatigue items. The scales are formatted on 1 to 4 pages for self-administration using a 5-point Likert rating scale (0 = Not at all; 1 = A little bit; 2 = Somewhat; 3 = Quite a Bit and 4 = Very much). Also, general health related quality of life (HRQoL), the FACT-An measures the impact of fatigue and other anemia-related symptoms on patient functioning and is used to assess the effect of treatments in various therapeutic areas, including MDS.
Mean Change in Quality of life measured with the EQ5D5L (European Quality of Life Five Dimension) scores | Baseline to 0-3 days prior to surgery and at 23-33 days postoperative
  Health-related quality of life will be measured using the EuroQol Five Dimensions (EQ-5D). The EQ-5D-5L is a valid extension of the 3-level questionnaire. It can be defined as a standardized non-disease specific value-based instrument to describe and value health-related quality of life. The instrument consists of two components: the EQ-5D descriptive system and the EQ visual analogue scale (EQ-VAS).The first part consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response categories (no problems, slight problems, moderate problems, severe problems, and extreme problems), from which a single EQ-5D index score can be calculated ranging from 0 (dead) to 1 (perfect health). The EQ-VAS measures one's self-perceived health today on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health) on which participants have to indicate their current health.
Mean Change in Quality of life measured with the SF-36 scores | Baseline to 0-3 days prior to surgery and at 23-33 days postoperative
  The SF-36 is a 36-item survey of health and well-being. The scale consists of eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health.
  Minimum Value: 0 (worst outcome) Maximum Value: 100 (best outcome)
Clinical surgical site infection | within 28 days following surgery
  Rate of participants presenting with clinical surgical site infection will be measured post-operation.
Clinical surgical complications | within 28 days following surgery
  Proportion of participants experiencing any complication post-operatively
Postoperative length of hospital stay | From Surgery date up to 60 days post surgery
  Mean and median length of stay (in days) in hospital following surgery
Rate of hospital readmission | from discharge date to 28 days post surgery
  Proportion of participants requiring re-admission to hospital following surgery after initial discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bisch SP, Woo L, Ljungqvist O, Nelson G. Ferric derisomaltose and Outcomes in the Recovery of Gynecologic oncology: ERAS (Enhanced Recovery After Surgery) (FORGE) - a protocol for a pilot randomised double-blinded parallel-group placebo-controlled study of the feasibility and efficacy of intravenous ferric derisomaltose to correct preoperative iron-deficiency anaemia in patients undergoing gynaecological oncology surgery. BMJ Open. 2023 Nov 9;13(11):e074649. doi: 10.1136/bmjopen-2023-074649. PMID 37945297